CLINICAL TRIAL: NCT01940874
Title: Cerebral Oxymetry at Elective Coronary and Valve Surgery: An Observational Study Using Norepinephrine to Maintain Arterial Blood Pressure on Cardio Pulmonary Bypass.
Brief Title: Cerebral Oxymetry at Elective Coronary and Valve Surgery.
Acronym: Co-HLM
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/823
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Coronary Artery Disease.; Aortic Valve Stenosis.; Aortic Valve Regurgitation.
Keywords: Cerebral Oximetry.; Aortic valve stenosis.; Aortic valve regurgitation.; Coronary artery disease.
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cerebral oximetry

SUMMARY:
Use of vasopressor to maintain Mean Arterial Pressure on Cardio Pulmonary Bypass can lead to decreased cerebral flow and oxygenation in individual patients and this can be detected by means of cerebral oxymetry.

ELIGIBILITY:
Inclusion Criteria:

* Patient age under 80.
* Patients should undergo elective coronary artery bypass grafting surgery (ACB) or heart valve surgery (AVR or MVR).
* The patient must be admitted at least 18 years of years.

Exclusion Criteria:

* Damage to the frontal lobes corresponding to the area where SCO2 monitored.
* Patients in pharmacological studies.
* Patients with known intracranial vascular anomalies or cerebral aneurysms.
* Patients with known neurological disease.
* Patients with known undergone cerebral insult, TIA or carotid stenosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We want to include 50 patients, both women and men, undergo elective coronary bypass surgery or valve surgeon in CPB with moderate hypothermia.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2011-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Cerebral oxymetry values | March 2013

CONTACTS AND LOCATIONS:
Overall Officials: Ove A. Hagen, MD, Principal Investigator — Oslo Ùniversity Hospital
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway